CLINICAL TRIAL: NCT00662714
Title: Open Randomised Prospective Comparative Multi-centre Intervention Study of Patients With Cystic Fibrosis and Early Diagnosed Diabetes Mellitus
Brief Title: Early Diagnosis of Diabetes Mellitus in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mukoviszidose Institut gGmbH (Other)
Collaborators: Novo Nordisk A/S (Industry); Mucoviscidose-ABCF2 (Unknown); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F01/01 CF-RD
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Cystic Fibrosis; Diabetes Mellitus
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus | interventions — repaglinide; Insulin, Short-Acting; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Repaglinide; oral
  Interventions: Drug: Repaglinide
- 2 (Active Comparator): short-acting Insulin (Actrapid)
  Interventions: Drug: short-acting Insulin (Actrapid)

INTERVENTIONS:
Drug: Repaglinide — oral; initial dose: 3x 0.5mg/d; 2 years
  Arms: 1
Drug: short-acting Insulin (Actrapid) — initial dose: 3x 0.05E/kg/d, injected; 2 years
  Other Names: Actrapid
  Arms: 2

SUMMARY:
Is oral therapy with Repaglinide equivalent to insulin therapy with three daily injections with respect to blood glucose control, weight and pulmonary function over 2 years in patients with cystic fibrosis and secondary diabetes mellitus? That is the question examined in the phase III trial.

DETAILED DESCRIPTION:
Diabetes mellitus may be present in patients with cystic fibrosis (mucoviscidosis) starting in the second decade of life. The prevalence increases rapidly with increasing age. As life-expectancy increases in CF, CF-related diabetes will be diagnosed more frequently in the future. Negative consequences of secondary diabetes in cystic fibrosis include:

* Catabolic metabolism
* Weight loss
* More frequent / more severe infections
* Deterioration of pulmonary function
* Reduced life-expectancy
* Diabetic micro vascular complications (retinopathy, nephropathy, neuropathy)

Up to date, no data are available to answer the question, whether secondary diabetes in CF should always be treated by insulin therapy. Several centres report the successful management of CF-related diabetes using oral anti-diabetic drugs at least for some years. Oral therapies would be less invasive for a patient group which is highly traumatised by a very demanding therapy (multiple drugs including antibiotics, pancreas enzymes, bronchodilators, mucolysis, in addition to physiotherapy, regular inpatient iv-antibiotic therapy etc, finally lung transplants in a subgroup of patients).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for the Screening:

* Diagnosed cystic fibrosis
* Age 10 years and older

Inclusion Criteria for the therapeutic part of the study:

* Newly diagnosed Diabetes mellitus in the screening

Exclusion Criteria:

Exclusion Criteria for Screening:

* Diabetic keto-acidosis (blood glucose > 350 mg/dl and arterial pH < 7.25)
* Already treated Diabetes mellitus by oral antidiabetic medication or insulin

Exclusion Criteria for the therapeutic part of the study:

* Systemic steroid therapy during the last 3 months
* Transplantation (status post TX or on the waiting list for TX)
* Beginning pulmonary insufficiency, FEV1 < 35% at pulmonary function test in stable condition
* Pregnancy
* Already diagnosed and treated diabetes mellitus
* Patients with diabetic keto-acidosis (blood glucose > 350 mg/dl and arterial pH < 7.25) with or without diabetic coma
* Severe liver insufficiency (chronic hepatitis B, AST or ALT twice the upper limit of normal, Quick's value < 70% which is a contraindication to use Repaglinide)
* Treatment with an indispensable important drug which contraindicates Repaglinide
* PEG/ gastric tube/ total parenteral alimentation for more than 4 weeks during the study
* CF-patients with type 1 diabetes
* Not patient's consent to randomisation and therapeutic trial
* Participation on other medical trial

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2001-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Ballmann, Prof. Dr., Principal Investigator — St. Josef Hospital,Alexandrinenstrasse 5,44791 Bochum, Germany; Reinhard Holl, Prof., Principal Investigator — Zentralinstitut für Biomedizinische Technik Ulm
Locations (36):
- Austria (2):
  - Universitätsklinik für Kinder- und Jugendheilkunde, Graz
  - Universitätsklinik für Kinder- und Jugendheilkunde, Vienna
- France (6):
  - CRCM adultes, Lille
  - CRCM adultes, Centre Hospitalier Lyon Sud, Lyon
  - APHP, CRCM pediatrique, Hopital Necker, Paris
  - APHP, CRCM pediatrique, Hopital Robert Debre, Paris
  - APHP, CRCM pediatrique, Hopital Cochin, Paris
  - CRCM adultes, Hopital Civil, Strasbourg
- Germany (27):
  - Helios Klinikum Emil von Behring, Berlin
  - Heliosklinikum Berlin-Buch, Berlin
  - Prof.-Hess-Kinderklinik/ Zentralkrankenhaus, Bremen
  - Zentralkrankenhaus "Links der Weser", Bremen
  - Klinik und Poliklinik für allgemeine Kinderheilkunde, Cologne
  - Universitätskinderklinik Düsseldorf, Düsseldorf
  - Klinik für Kinder und Jugendliche Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Ruhrlandklinik Essen, Essen
  - Zentrum für Kinderheilkunde Frankfurt, Frankfurt
  - Med. Klinik II, Allergologie und Pneumologie, Frankfurt
  - Klinik Schillerhöhe, Gerlingen
  - Klinik und Poliklinik für Kinder- und Jugendmedizin, Greifswald
  - Altona - Klinik, Hamburg
  - Medizinische Hochschule Hannover, Abt. Kinderheilkunde, Hanover
  - Medizinische Hochschule Hannover, CF-Ambulanz f. Erwachsene, Hanover
  - Klikum der Universität Heidelberg, Kinderklinik, Heidelberg
  - Universitätsklinik für Kinder- und Jugendmedizin, Homburg
  - Kinderkrankenhaus Park Schönfeld, Kassel
  - Städtisches Krankenhaus Kiel, Kiel
  - Universitätsklinik Mainz, Mainz
  - Clemenshospital, Münster
  - Elisabeth Kinderkrankenhaus, Oldenburg
  - Kinderhospital Osnabrück, Osnabrück
  - Kinderklinik Dritter Orden, Sozialpädiatrisches Zentrum, Passau
  - Universitätsklinik für Kinder- und Jugendmedizin, Tübingen
  - Julius-Maximilians Universität, Kinderpoliklinik, Würzburg
- Centro Fibrosi Cistica, Verona, Italy

REFERENCES:
- [Derived] Onady GM, Stolfi A. Drug treatments for managing cystic fibrosis-related diabetes. Cochrane Database Syst Rev. 2020 Oct 19;10(10):CD004730. doi: 10.1002/14651858.CD004730.pub5. PMID 33075159
- [Derived] Ballmann M, Hubert D, Assael BM, Staab D, Hebestreit A, Naehrlich L, Nickolay T, Prinz N, Holl RW; CFRD Study Group. Repaglinide versus insulin for newly diagnosed diabetes in patients with cystic fibrosis: a multicentre, open-label, randomised trial. Lancet Diabetes Endocrinol. 2018 Feb;6(2):114-121. doi: 10.1016/S2213-8587(17)30400-X. Epub 2017 Dec 5. PMID 29199116
- [Derived] Ballmann M, Hubert D, Assael BM, Kronfeld K, Honer M, Holl RW; CFRD Study group. Open randomised prospective comparative multi-centre intervention study of patients with cystic fibrosis and early diagnosed diabetes mellitus. BMC Pediatr. 2014 Mar 11;14:70. doi: 10.1186/1471-2431-14-70. PMID 24620855
- [Derived] Schmid K, Fink K, Holl RW, Hebestreit H, Ballmann M. Predictors for future cystic fibrosis-related diabetes by oral glucose tolerance test. J Cyst Fibros. 2014 Jan;13(1):80-5. doi: 10.1016/j.jcf.2013.06.001. Epub 2013 Jun 25. PMID 23809507